CLINICAL TRIAL: NCT00837018
Title: Exercise Intolerance in Obstructive Sleep Apnea Syndrome Patients: Cardiovascular and Metabolic Characterisation During Exercise. Treatments Effect.
Brief Title: Exercise Intolerance in Obstructive Sleep Apnea Syndrome Patients
Acronym: EXAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 0520; DGS 2005/0312 (Registry Identifier: DGS)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSAS; exercise; metabolic; cardio-vascular
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical exercise program (Experimental): 45 min, 3 times a week
  Interventions: Other: physical exercise program

INTERVENTIONS:
Other: physical exercise program — 45 min, 3times a week

SUMMARY:
The syndrome of obstructive sleep apnea (OSAS) is a public health problem that affects 2 to 4% of the general population. The patients with OSAS frequently complain of intolerance to exercise muscle fatigue and a significant even if they have not been fully characterized in the literature.

The anomalies in the exercise of patients with OSAS could be due to metabolic changes (insulin resistance and oxidative stress) and cardiovascular (impaired vascular reactivity).

Our goal is both to determine whether these anomalies exist in patients with OSAS not obese, consider their relationship with the alteration of exercise capacity, and their reversibility in conventional PPC or by using the effects of physical activity regular.In this study Objectives: To establish whether the metabolic and vascular abnormalities associated with OSAS are associated with decreased parameters of physical fitness in relation to witnesses matched for age, sex and body mass index. Determine the effects of a re-training exercise on these parameters compared to the reference treatment, continuous positive pressure.

Main objective: To compare the exercise capacity of OSAS patients compared with that of witnesses matched for age, sex and body mass index.

Secondary objectives: To compare the effect of conventional treatment by continuous positive pressure (CPP) on cardiovascular and metabolic abnormalities of OSAS, with a therapeutic modality most original, physical activity.

Methodology: Test physiopathological parallel group, controlled, randomized.

DETAILED DESCRIPTION:
Study type : Physiopathology trial Study design : Prospective randomized controled trial

Expected Total Enrollment : 45 patients + 15 control subjects

Tested treatment : Physical exercise program (45 minutes, 3 times a week) Reference treatment : continuous positive airway pressure Treatment duration : 12 weeks (3 months) Total study duration : 2 years

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study : 18 Years and above
* Genders Eligible for Study: Both
* Non obese : body mass index (BMI < 30 kg/m2)
* Sedentary subjects : less physical activity than 30 minutes 3 time a week
* and VOORIPS physical activity level questionnaire score < 9.

Obstructive sleep apnea syndrome (OSAS) patients :

* Recently diagnosed (< 3 months)
* AHI > 30 / hour (polysomnographic monitoring measurement)

Exclusion Criteria:

* Excessive daytime sleepiness (Epworth score > 12)
* Cardiovascular pathology (except controlled hypertension)
* Pathology interacting with physical activity
* Diabetes (known or treated)
* Other participation to a clinical trial at the same

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Comparison of maximal oxygen consumption : OSAS patient versus control subjects. | when the last patient realised the last visit

SECONDARY OUTCOMES:
To compare physical exercise program to continuous positive airway pressure after 12 weeks of treatment in OSAS patients. | when the last patient realised the last visit

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, doctor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU, medecine du sport, Grenoble, France